CLINICAL TRIAL: NCT04448977
Title: A Biomarker for Cognitive Fatigue Using Functional Imaging in MS
Brief Title: Examining Effects of Ocrevus on Cognitive Fatigue Using fMRI
Status: Recruiting | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: R-1104-20
Record Dates: First submitted 2020-06-15; First posted 2020-06-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; cognitive fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Multiple Sclerosis group 1: Individuals with Multiple Sclerosis who are going to be starting Ocrevus as determined by Neurologist as part of clinical care.
  Interventions: Drug: Ocrevus
- Multiple Sclerosis group 2: Individuals with Multiple Sclerosis who are going to be starting Copaxone as determined by Neurologist as part of clinical care.
- Healthy Controls: Healthy individuals who are age, gender and education matched to the other groups.

INTERVENTIONS:
Drug: Ocrevus — Participants with MS will be divided into two treatment groups: those who will begin to take Ocrevus (the "early Ocrevus" group (EO), and those who plan to be begin treatment with Glatimer acetate SC (Copaxone) (EC). Both groups will be matched to the EO group for age, gender and education. The HC group will be free of neurological disease or injury and will be matched to the EO group for age, gender, and education.
  Groups: Multiple Sclerosis group 1

SUMMARY:
The purpose of this research study is to investigate the effectiveness of MS Disease modifying medications on cognitive fatigue in persons with relapsing remitting multiple sclerosis (RRMS). Cognitive fatigue is the kind of fatigue that occurs after intense mental concentration as after a session of problem solving.

DETAILED DESCRIPTION:
The researchers aim is to investigate the effects of disease modifying treatments on cognitive fatigue and on specific brain areas that have been shown to underlie cognitive fatigue in individuals with Multiple Sclerosis (MS). The researchers will investigate the effects on the cognitive fatigue that develops during the performance of a demanding task, and also on how cognitive fatigue changes as a function of duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64.
* Relapsing remitting multiple sclerosis
* Been newly prescribed a new disease modifying medication for MS (either Ocrevus or Copaxone)
* or healthy volunteer who can speak English fluently.

Exclusion Criteria:

* History of head injury, stroke, seizures, or any other significant neurological event other than MS
* Flare up of MS symptoms within the past month.
* History of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder.
* Pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* left handed.
* Not able to have an MRI

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who have Relapsing remitting Multiple Sclerosis and Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain activation (BOLD signal) | Measured for change at 3 time points (before, six months and 12 months after intervention)
  A change in brain activation as measured with functional magnetic resonance imaging through blood oxygen level dependent signal will be measured in association with cognitive fatigue (as measured by the Visual Analogue scale during performance of the modified Symbol Digit Modality and Modified Fatigue Impact Scale).

SECONDARY OUTCOMES:
Fatigue onset | Measured for change at 3 time points for change (before, six months and 12 months after intervention)
  A change in the speed with which modified Symbol Digit Modality task (a cognitively demanding task) induces fatigue in MS (as measured by the Visual Analogue scale and Modified Fatigue Impact Scale).

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No